CLINICAL TRIAL: NCT04820738
Title: Effects of Sensory Motor Training on Balance and Proprioception Among Post-Menopausal Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2050 Sehar Shabeer
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Post Menopaused Female
Keywords: Postmenopausal, Obese, Balance, Proprioception
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Sensorimotor training exercises include wall slides , core exercises (Planks, leg raises, crunches, bridging) balance exercises (single leg side lift, leg lift with dumble, balance on stability ball) on unstable surface for 50-60 min (3 sets of 10 rep) of exercises and gait training (different patterns of walking).
  Interventions: Other: Sensorimotor training exercises
- Control group (Active Comparator): Cut back on high-fat foods. Drink plenty of water Use sugar and salt in moderation. Eat fruits and vegetables Get enough calcium Pump up your iron. Get enough fiber
  Interventions: Other: Without Sensorimotor training exercises

INTERVENTIONS:
Other: Sensorimotor training exercises — Sensorimotor training exercises include wall slides , core exercises (Planks, leg raises, crunches, bridging) balance exercises (single leg side lift, leg lift with dumble, balance on stability ball) on unstable surface for 50-60 min (3 sets of 10 rep) of exercises and gait training (different patterns of walking
  Arms: Experimental group
Other: Without Sensorimotor training exercises — Cut back on high-fat foods. Drink plenty of water Use sugar and salt in moderation. Eat fruits and vegetables Get enough calcium Pump up your iron. Get enough fiber
  Arms: Control group

SUMMARY:
Postmenopausal obese women often have difficulties with balance and proprioception. Sensorimotor training is an important part of physical therapy interventions, with emerging evidence that it could be beneficial for postmenopausal obese women.

Objective: To find the impact of sensorimotor training on balance and proprioception among postmenopausal obese women.

DETAILED DESCRIPTION:
Randomized clinical trial was conducted on postmenopausal obese women population with impaired balance and proprioception on inclusion & exclusion criteria, sample size of 40, ages ranged from 45 to 65 years included. Group A received SMT and Group B received CT. The interval of treatment was 6 weeks. Data is collected from THQ Samundri. FRT, TUG, OLS utilized to assess the pre-and post-estimations of postural strength.

ELIGIBILITY:
Inclusion Criteria:

* • Post-menopausal obese women

  * BMI ≥30
  * Participants independent in ADLs
  * self-ambulatory
  * healthy (having no known condition in which sensorimotor exercises would be contraindicated.)

Exclusion Criteria:

* • History of ankle sprain

  * Uncontrolled diabetes mullites
  * Presence of orthopaedic problems.
  * Neurological disorders.
  * Psychological problems.
  * Cognitive issues.
  * People with severe visual issues

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — post manupausal women obesty BMI More than 30
Enrollment: 44 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Functional Reach Test (FRT) | 2 months
  Functional Reach Test (FRT) is a clinical outcome measure used to asses dynamic balance in one simple task.
Time Up and Go Test (TUG) | 2 months
  Time Up and Go test is used to assess the individual's mobility, static and dynamic balance walking ability and risk of fall among older adults. Intratester and intertester reliability (ICC) in elderly populations
One Leg Stance Test (OLS) | 2 months
  The Single leg Stance (SLS) Test is used to evaluate static postural and balance control with one eye open and standing on one leg

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabrera-Martos I, Jimenez-Martin AT, Lopez-Lopez L, Rodriguez-Torres J, Ortiz-Rubio A, Valenza MC. Effects of a core stabilization training program on balance ability in persons with Parkinson's disease: a randomized controlled trial. Clin Rehabil. 2020 Jun;34(6):764-772. doi: 10.1177/0269215520918631. Epub 2020 Apr 29. PMID 32349543
- [Background] Marsden JF. Cerebellar ataxia. Handb Clin Neurol. 2018;159:261-281. doi: 10.1016/B978-0-444-63916-5.00017-3. PMID 30482319
- [Background] Yang WC, Wang HK, Wu RM, Lo CS, Lin KH. Home-based virtual reality balance training and conventional balance training in Parkinson's disease: A randomized controlled trial. J Formos Med Assoc. 2016 Sep;115(9):734-43. doi: 10.1016/j.jfma.2015.07.012. Epub 2015 Aug 13. PMID 26279172
- [Background] Silva PB, Oliveira AS, Mrachacz-Kersting N, Kersting UG. Effects of wobble board training on single-leg landing neuromechanics. Scand J Med Sci Sports. 2018 Mar;28(3):972-982. doi: 10.1111/sms.13027. Epub 2018 Jan 30. PMID 29193314
- [Background] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Background] Skards IaV, Vitols AV, Matisone DR, Dzerve-Talums VIa, Skarda IIa. [Correlation of functional and structural changes of the cardiovascular system in hypertensive disease]. Fiziol Zh SSSR Im I M Sechenova. 1988 Nov;74(11):1628-35. Russian. PMID 2977590
- [Background] Geiger M, Supiot A, Zory R, Aegerter P, Pradon D, Roche N. The effect of transcranial direct current stimulation (tDCS) on locomotion and balance in patients with chronic stroke: study protocol for a randomised controlled trial. Trials. 2017 Oct 23;18(1):492. doi: 10.1186/s13063-017-2219-6. PMID 29061169
- [Background] Martins E Silva DC, Bastos VH, de Oliveira Sanchez M, Nunes MK, Orsini M, Ribeiro P, Velasques B, Teixeira SS. Effects of vestibular rehabilitation in the elderly: a systematic review. Aging Clin Exp Res. 2016 Aug;28(4):599-606. doi: 10.1007/s40520-015-0479-0. Epub 2015 Oct 28. PMID 26511625
- [Background] Pellegrino L, Giannoni P, Marinelli L, Casadio M. Effects of continuous visual feedback during sitting balance training in chronic stroke survivors. J Neuroeng Rehabil. 2017 Oct 16;14(1):107. doi: 10.1186/s12984-017-0316-0. PMID 29037206
- [Background] Gomiero AB, Kayo A, Abraao M, Peccin MS, Grande AJ, Trevisani VF. Sensory-motor training versus resistance training among patients with knee osteoarthritis: randomized single-blind controlled trial. Sao Paulo Med J. 2018 Jan-Feb;136(1):44-50. doi: 10.1590/1516-3180.2017.0174100917. Epub 2017 Dec 7. PMID 29236934